CLINICAL TRIAL: NCT04056819
Title: A Phase I, Open Label Study to Evaluate the Safety and to Explore Efficacy of Allogeneic Umbilical Cord Mesenchymal Stem Cells in Patients with ST-elevation Acute Myocardial Infarction
Brief Title: Evaluate the Safety and Explore Efficacy of Umbilical Cord Mesenchymal Stem Cells in Acute Myocardial Infarction
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Ever Supreme Bio Technology Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ES-CMSC01-A1101
Record Dates: First submitted 2019-07-31; First posted 2019-08-14 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2022-03

CONDITIONS: Acute Myocardial Infarction

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- UMSC01 (Experimental): UMSC01 cells mixed with normal saline will be administered to patients after the onset of heart attack.
  Interventions: Biological: Allogeneic umbilical cord mesenchymal stem cells

INTERVENTIONS:
Biological: Allogeneic umbilical cord mesenchymal stem cells — UMSC01 cells will be one single IC infusion followed by one single IV infusion with 12 months of follow up after treatment.

SUMMARY:
This study is a first-in-human assessment of safety of using UCMSC in patients with AMI via a combination of IC and IV stem cell administration. The novelty of the current UMSC01 treatment study is the dual route of administration. Since dual administration of UCMSC via IC and IV had never been conducted in humans, there may be unknown risks to humans not predicted from the preclinical studies. However, the risk to patients in this trial will be minimized by rigorous adherence to the eligibility criteria, use of appropriate dose and concentration of stem cells, standardized techniques of stem cell infusion, and intensive patient monitoring during and after stem cell infusion.

DETAILED DESCRIPTION:
Cardiovascular disease is the leading cause of death in the developed world, with global deaths due to coronary artery disease estimated to increase from 7.3 million in 2008 to 25 million by 2020 WHO, 2011.

The leading symptom that initiates the diagnostic and therapeutic cascade in patients with suspected acute coronary syndromes (ACS) is chest pain.

Most patients will ultimately develop an ST elevation myocardial infarction (STEMI). The mainstay of treatment in these patients is immediate reperfusion by primary angioplasty or fibrinolytic therapy. Basically, STEMI comprises approximately 25% to 40% of myocardial infarction (MI) presentations. Acute STEMI is a major cause of morbidity, mortality, and disability.

This product is a new cell therapy product for treating AMI and produced by Ever Supreme Bio Technology Co., Ltd in Taiwan. For animal studies, UMSC01 has been demonstrated its effectiveness for AMI and stroke. The rats with coronary artery ligation receiving intravenous injection of UMSC01 showed significantly improved cardiac function.

ELIGIBILITY:
Donor-Inclusion Criteria:

1. Pregnant women who are aged ≥ 20, <50 years old on date of consent.
2. Pregnant women who are willing to and has given her signed written informed consent.
3. Pregnant women whose gestation age ≥ 34 weeks and have intact placenta.
4. Pregnant women who have not had any complication of pregnancy.
5. Pregnant women who are willing to provide a personal and family medical history (as much available) of herself and the biologic father (as much available), prior to or following collection of the umbilical cord.

Donor-Exclusion Criteria:

1. Pregnant women who have clinically severe and/or life-threatening disease(s) such as uncontrolled diabetes mellitus (fasting sugar level > 250 mg/dL) and malignant tumor.
2. Pregnant women who have been tested positive for the following tests within 7 days before or after umbilical cord acquirement:

   * Human immunodeficiency virus-1 (HIV-I): anti-HIV-I and nucleic acid test (NAT)
   * HIV-II
   * Hepatitis B virus (HBV): Hepatitis B surface antigen (HBsAg), anti- Hepatitis B core (HBc) and NAT
   * Hepatitis C virus (HCV): anti-HCV and NAT
   * Cytomegalovirus (CMV) (Note: If the pre-screened CMV result shows positive 8 weeks prior to umbilical cord acquirement will also be excluded.)
   * Treponema pallidum
   * Chlamydia trachomatis
   * Neisseria gonorrhea
   * Human T cell leukemia virus-I/II (HTLV-I/II)
   * West Nile virus (WNV) NAT
3. Pregnant women are with increased risk for Creutzfeldt-Jakob disease (CJD) if you have received a non-synthetic dura mater transplant, human pituitary-derived growth hormone, or have one or more blood relatives diagnosed with CJD.
4. Pregnant women had spent three months or more cumulatively in the United Kingdom from the beginning of 1980 through the end of 1996; or had received any transfusion of blood or blood components in the U.K. or France between 1980 and the present; or lived 5 years or more cumulatively in Europe.
5. Pregnant women or her sexual partners were born or lived in certain countries in Africa (Cameroon, Central African Republic, Chad, Congo, Equatorial Guinea, Gabon, Niger, or Nigeria) after 1977 (risk factor for HIV group O).
6. Pregnant women who have medical diagnosis of Zika virus (ZIKV) infection or residence in, or travel to, an area with active ZIKV transmission (according to the list from Centers for Disease Control and Prevention. Zika Virus: Areas with Zika.) at any point during that pregnancy.
7. Pregnant women who have sex at any point during that pregnancy with a male who is known to medical diagnosis of ZIKV infection or residence in, or travel to, an area with active ZIKV transmission.
8. Pregnant women who have received blood infusion or stayed for more than 3 months in WNV potential countries.
9. Pregnant women who have unexplained post-donation febrile illness with headache or other symptoms suggestive of WNV infection (i.e., flu-like symptoms that include fever with headache, eye pain, body aches, generalized weakness, new skin rash or swollen lymph nodes or other evidence of WNV infection) within two weeks.
10. Pregnant women who have medical history of tuberculosis.
11. Pregnant women who have medical history of malignant tumor.
12. Fetuses that have found with genetic disease in prenatal checkups.
13. Pregnant women who would like to store cord blood or umbilical cord cells, other than this study usage.
14. Pregnant women who are not suitable to donate as judged by the Investigator(s).

Subject-Inclusion Criteria:

1. Male or female patients are aged ≥20, <76 years old on date of consent.
2. Patients who presented typical ischemic chest pain within 12 h after symptoms onset and are diagnosed first acute STEMI according to the 2013 American College of Cardiology (ACC) Foundation/American Heart Association (AHA) guideline for the Management of STEMI.
3. Patients who have undergone standard-of-care for STEMI; the immediate reperfusion management should include primary percutaneous coronary intervention (PCI), aspiration thrombectomy and adjunctive antithrombotic therapy within 12 hours after the onset of symptoms.
4. Patients who undergo successful acute reperfusion therapy (residual stenosis visually <50% and TIMI flow ≥2) with placement of an intracoronary stent have a patent infarct-related artery suitable for cell infusion to the target area of abnormal wall motion following myocardial infarction.
5. Patients who have left ventricular ejection fraction (LVEF) ≥ 30% and < 50% diagnosed by echocardiogram.
6. Patients are willing to sign informed consent or assent by the next of kin.
7. Patients who have stable vital signs for at least 48 hours, defined as normal respiration, afebrile, systolic pressure ≥ 90 mmHg and < 180 mmHg, heart rate > 50/min and <110/min.
8. Adequate pulmonary function test defined as a force expiratory volume 1s (FEV1) > 50% predicted and peripheral artery oxygen saturation ≥95% at room air.
9. All male patients and female patients with child-bearing potential (between puberty and 2 years after menopause) should use appropriate contraception method(s) shown below, for at least 4 weeks after UMSC01 treatment.

   1. Total abstinence (when this is in line with the preferred and usual lifestyle of the subject. Periodic abstinence (e.g., calendar, ovulation, symptothermal, post-ovulation methods) and withdrawal are not acceptable methods of contraception).
   2. Female sterilization (have had surgical bilateral oophorectomy with or without hysterectomy) or tubal ligation at least six weeks before taking study treatment. In case of oophorectomy alone, only when the reproductive status of the woman has been confirmed by follow up hormone level assessment.
   3. Male sterilization (at least 6 months prior to screening). For female subjects on the study, the vasectomized male partner should be the sole partner for that subject
   4. Combination of any two of the following listed methods: (d.1+d.2 or d.1+d.3, or d.2+d.3):

   d.1 Use of oral, injected or implanted hormonal methods of contraception or other forms of hormonal contraception that have comparable efficacy (failure rate <1%), for example hormone vaginal ring or transdermal hormone contraception.

   d.2 Placement of an intrauterine device (IUD) or intrauterine system (IUS). d.3 Barrier methods of contraception: Condom or Occlusive cap (diaphragm or cervical/vault caps) with spermicidal foam/gel/film/cream/vaginal suppository.

Subject-Exclusion Criteria:

1. Patients with cardiogenic shock (defined as systolic blood pressure < 80 mmHg requiring vasopressors, intra-aortic balloon pump (IABP) or extracorporeal membrane oxygenation (ECMO).
2. Patients who have severe aortic stenosis or regurgitation according to the recommendation of the 2014 ACC/AHA guideline for the Management of Patients with Valvular Heart Disease.
3. Patients who have severe mitral stenosis or regurgitation according to the recommendation of 2014 ACC/AHA guideline for the Management of Patients with Valvular Heart Disease.
4. Patients who need to undergo staged coronary intervention therapy or coronary artery bypass grafting (CABG) surgery.
5. Patients who have immuno-compromised condition, or is with known clinically significantly autoimmune conditions or is receiving immunosuppressive treatments.
6. Patients who are unable to undergo cardiac magnetic resonance imaging (CMRI) scans for any reason.
7. Patients with inadequate hepatic and renal function after onset of STEMI: Aspartate aminotransferase (AST) and Alanine aminotransferase (ALT) ≥ 4 x upper limit of normal (ULN); estimated glomerular filtration rate (eGFR) < 30 mL/min.
8. For patients with diabetes mellitus: patients with uncontrolled diabetes mellitus (fasting sugar level > 250 mg/dL).
9. Patients who have medical history of malignant tumor or other clinically significant cardiovascular diseases that will confound the evaluation of this study.
10. Patients who participated other clinical trial within last 3 months.
11. Female patient who is pregnant, lactating or with child-bearing potential but not practicing effective contraceptive method(s).
12. Patients not suitable to participate the trial as judged by the Investigator(s).

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2019-05-27 (Actual); Primary Completion 2021-08-02 (Actual); Study Completion 2021-12-17 (Actual)

PRIMARY OUTCOMES:
Incidence of Treatment emergent adverse event (TEAE) as presented by MedDRA coding system | from visit 2 to 12-month follow-up period
  TEAE incidences over the study period
Incidence of Serious adverse event (SAE) as presented by MedDRA coding system | from visit 2 to 12-month follow-up period
  SAE incidences over the study period
Incidence of Suspected and unexpected serious adverse reaction (SUSAR) as presented by MedDRA coding system | from visit 2 to 12-month follow-up period
  SUSAR incidences over the study period

SECONDARY OUTCOMES:
New York Heart Association (NYHA) Classification | 12 weeks
  The NYHA classification is used to grade the severity of functional limitations in a patient with heart failure with Class I=no limitations to Class IV=unable to carry on any physical activity without discomfort.
Incidence of major adverse cardiovascular events (MACE) | from screen visit to 12-month follow-up period
  MACE are defined as death, recurrent MI, stroke, target vessel revascularization.
Serum level of amino-terminal pro-brain natriuretic peptide (NT pro-BNP) | 52 weeks
  Change of serum level of NT pro-BNP from baseline visit to subsequent visits will be summarized by descriptive statistics.
Pulmonary function test | 52 weeks
  The FEV1 will be tested by Spirometry and recorded.
Echocardiogram | 52 weeks
  Change of regional left ventricular wall motion score in total score from baseline visit to subsequent visits will be displayed by descriptive statistics
Echocardiogram | 52 weeks
  Change of LVESV in mL from baseline visit to subsequent visits will be displayed by descriptive statistics
Echocardiogram | 52 weeks
  Change of LVEDV in mL from baseline visit to subsequent visits will be displayed by descriptive statistics
Echocardiogram | 52 weeks
  Change of LV fractional shortening in % from baseline visit to subsequent visits will be displayed by descriptive statistics
Echocardiogram | 52 weeks
  Change of LVEF in % from baseline visit to subsequent visits will be displayed by descriptive statistics
Cardiac MRI (cMRI) for baseline and efficacy evaluation | 52 weeks
  Change of LVEF in % from baseline visit to subsequent visits will be summarized by descriptive statistics
Cardiac MRI (cMRI) for baseline and efficacy evaluation | 52 weeks
  Change of regional left ventricular wall motion score in total score from baseline visit to subsequent visits will be summarized by descriptive statistics
Cardiac MRI (cMRI) for baseline and efficacy evaluation | 52 weeks
  Change of LVESV in mL from baseline visit to subsequent visits will be summarized by descriptive statistics
Cardiac MRI (cMRI) for baseline and efficacy evaluation | 52 weeks
  Change of LVEDV in mL from baseline visit to subsequent visits will be summarized by descriptive statistics
Cardiac MRI (cMRI) for baseline and efficacy evaluation | 52 weeks
  Change of scar volume in % from baseline visit to subsequent visits will be summarized by descriptive statistics
Cardiac MRI (cMRI) for baseline and efficacy evaluation | 52 weeks
  Change of myocardial fibrosis quantification in % from baseline visit to subsequent visits will be summarized by descriptive statistics

OTHER OUTCOMES:
Cardiac Positron emission tomography (CPET) to demonstrate perfusion-metabolism mismatch | 52 weeks
  The change of myocardial perfusion (17 segment bull's eye polar plot) from baseline to subsequent visits will be summarized by descriptive statistics. In addition, the interpretation of CPET results will be provided by the investigator in narrative form and will be listed in a listing.
Tl-201 single photon emission computed tomography (SPECT) scan to determine myocardial infarction occurrence | 52 weeks
  The change of myocardial perfusion (17 segment bull's eye polar plot) from baseline to subsequent visits will be summarized by descriptive statistics. In addition, the interpretation of SPECT results will be provided by the investigator in narrative form and will be listed in a listing.

CONTACTS AND LOCATIONS:
Overall Officials: Woei Shyu, Study Director — Ever Supreme Bio Technology Co., Ltd.
Locations (1):
- China Medical University Hospital, Taichung, Non-US, Taiwan

REFERENCES:
- [Background] Hsiao LC, Lin YN, Shyu WC, Ho M, Lu CR, Chang SS, Wang YC, Chen JY, Lu SY, Wu MY, Li KY, Lin YK, Tseng WI, Su MY, Hsu CT, Tsai CK, Chiu LT, Chen CL, Lin CL, Hu KC, Cho DY, Tsai CH, Chang KC, Jeng LB. First-in-human pilot trial of combined intracoronary and intravenous mesenchymal stem cell therapy in acute myocardial infarction. Front Cardiovasc Med. 2022 Aug 9;9:961920. doi: 10.3389/fcvm.2022.961920. eCollection 2022. PMID 36017096
- See also: First-in-human pilot trial of combined intracoronary and intravenous mesenchymal stem cell therapy in acute myocardial infarction — https://www.frontiersin.org/articles/10.3389/fcvm.2022.961920/full